CLINICAL TRIAL: NCT03792477
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 2-TREATMENT SINGLE-DOSE, CROSS-OVER STUDY, 2-PART DESIGN TO EVALUATE THE BIOEQUIVALENCE AND TOLERABILITY OF TESTOSTERONE CYPIONATE FOLLOWING INTRAMUSCULAR (IM) INJECTION IN HEALTHY HYPOGONADAL MALE SUBJECTS
Brief Title: A Bioequivalence Study of Testosterone Cypionate in Hypogonadal Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B5341002; DEPO-T BE STUDY (Other: Alias Study Number)
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, 2-treatment, 2-period, single dose (200 mg), cross-over study, 2-part design to evaluate the bioequivalence and tolerability of a reformulated presentation of testosterone cypionate relative to a currently marketed and approved formulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Treatment A (Experimental): Single 200mg IM testosterone cypionate solution (Test formulation)
  Interventions: Biological: Test formulation
- Part 1: Treatment B (Active Comparator): Single 200 mg IM testosterone cypionate solution (Reference formulation)
  Interventions: Biological: Reference formulation
- Part 2: Treatment A (Experimental): Single 200 mg IM testosterone cypionate solution (Test formulation)
  Interventions: Biological: Test formulation
- Part 2: Treatment B (Active Comparator): Single 200 mg IM testosterone cypionate solution (Reference formulation)
  Interventions: Biological: Reference formulation

INTERVENTIONS:
Biological: Test formulation — A single testosterone cypionate solution for injection (new formulation) 200 mg dose administered IM deep in the gluteal muscle (Test formulation).
  Arms: Part 1: Treatment A; Part 2: Treatment A
Biological: Reference formulation — A single testosterone cypionate solution for injection (currently marketed formulation) 200 mg dose administered IM deep in the gluteal muscle (Reference formulation).
  Arms: Part 1: Treatment B; Part 2: Treatment B

SUMMARY:
This is an open-label, 2-treatment, 2-period, single dose (200 mg, IM) cross-over study, 2-part design to evaluate the bioequivalence (BE) of a reformulated presentation (test) of testosterone cypionate solution for injection relative to the currently approved marked formulation (reference). In the first part of the study (Part 1), an estimate of the exposure variability will be evaluated for both test and reference. This will help guide sample size in Part 2. Part 2 will be powered to assess the BE of both test and reference formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Hypogonadal male subjects who, at the time of screening, are otherwise healthy and between the ages of 18 and 65 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12 lead electrocardiogram (ECG), or clinical laboratory tests.

   Hypogonadism is defined as serum testosterone levels below 2.5 ng/mL (250 ng/dL).
2. Body mass index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lb).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Subjects who are currently being treated for hypogonadism. This is defined as either patients who have received a testosterone injectable product within the past 3 months or have used a transdermal or gel product within the past 2 weeks.
3. A positive urine drug test.
4. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
6. Screening supine BP greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
7. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
8. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level greater than or equal to 3 times the upper limit of normal (ULN).
   * Total bilirubin level greater than or equal to 1.5 times the ULN; subject with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is less than or equal to ULN.
9. Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol [Contraception (Section 4.3.4)] for the duration of the study and for at least 45 days after the last dose of investigational product.
10. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of greater than or equal to 1 g/day. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
12. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
13. History of sensitivity to heparin or heparin induced thrombocytopenia.
14. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
15. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
16. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
17. Subjects with carcinoma of the breast.
18. Subjects with known or suspected carcinoma of the prostate gland.
19. Subjects who are hypersensitive to testosterone cypionate or its inactive ingredients.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Avail Clinical Research, DeLand, Florida
  - Syneos Health, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5341002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 parts in the study, different participants were enrolled into the 2 individual parts.
Pre-assignment Details: This study was a multi-period crossover study. In Part 1, there were 2 treatment periods with a washout period of 45 days. In Part 2, there were 3 treatment periods with 2 washout periods of 45 days each.
Groups:
- Part 1: Treatment A>Treatment B: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (intramuscular [IM]) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This is the Part 1 Sequence 1, where participants received the treatments in the order of A, B.
- Part 1: Treatment B>Treatment A: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This is the Part 1 Sequence 2, where participants received the treatments in the order of B, A.
- Part 2: Treatment A>Treatment B>Treatment B: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This is the Part 2 Sequence 1, where participants received the treatments in the order of A, B, B.
- Part 2: Treatment B>Treatment A>Treatment B: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This is the Part 2 Sequence 2, where participants received the treatments in the order of B, A, B.
- Part 2: Treatment B>Treatment B>Treatment A: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This is the Part 2 Sequence 3, where participants received the treatments in the order of B, B, A.
Period: Overall Study
Arm/Group | Part 1: Treatment A>Treatment B | Part 1: Treatment B>Treatment A | Part 2: Treatment A>Treatment B>Treatment B | Part 2: Treatment B>Treatment A>Treatment B | Part 2: Treatment B>Treatment B>Treatment A
Started | 6 | 6 | 21 | 21 | 20
Completed | 6 | 6 | 19 | 20 | 19
Not Completed | 0 | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- Part 1: Treatment A>Treatment B: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This is the Part 1 Sequence 1, where participants received the treatments in the order of A, B.
- Total: Total of all reporting groups
Arm/Group | Part 1: Treatment A>Treatment B | Part 1: Treatment B>Treatment A | Part 2: Treatment A>Treatment B>Treatment B | Part 2: Treatment B>Treatment A>Treatment B | Part 2: Treatment B>Treatment B>Treatment A | Total
Number analyzed (Participants) | 6 | 6 | 21 | 21 | 20 | 74
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0 | 0 | 0 | 0 | 0 | 0
  18-45 Years | 0 | 0 | 4 | 3 | 5 | 12
  45-65 Years | 6 | 6 | 17 | 18 | 15 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 21 | 21 | 20 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 18 | 18 | 17 | 64
  Black or African American | 0 | 1 | 3 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Corrected Area Under The Serum Concentration-time Profile From Time 0 to The Last Quantifiable Concentration (AUClast) of Total Testosterone (Part 1).
Description: The AUClast of total testosterone in Part 1 of the study was observed directly from data. The baseline endogenous testosterone level was the mean of the 4 predose PK samples, an average baseline correction of endogenous total testosterone levels was calculated.
Time Frame: At -1, -0.5, -0.25, 0 hours predose and at 1, 8, 24, 36, 48, 72, 96, 120, 144, 168, 240, 336 and 480 hours postdose.
Population: The analysis population included all participants randomized and treated who had at least 1 of the pharmacokinetic parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Treatment A; Treatment B: This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 1444 (62) | 1362 (47)

2. Primary Outcome: Corrected AUC From Tme 0 Extrapolated to Infinite Time (AUCinf) of Total Testosterone (Part 1).
Description: The AUCinf of total testosterone in Part 1 of the study was observed directly from data. The baseline endogenous testosterone level was the mean of the 4 predose PK samples, an average baseline correction of endogenous total testosterone levels was calculated.
Time Frame: At -1, -0.5, -0.25, 0 hours predose and at 1, 8, 24, 36, 48, 72, 96, 120, 144, 168, 240, 336 and 480 hours postdose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 9 | 10
ng*hr/mL | 1424 (66) | 1392 (41)

3. Primary Outcome: Corrected Maximum Observed Concentration (Cmax) of Total Testosterone (Part 1).
Description: The Cmax of total testosterone in Part 1 of the study was observed directly from data. The baseline endogenous testosterone level was the mean of the 4 predose PK samples, an average baseline correction of endogenous total testosterone levels was calculated.
Time Frame: At -1, -0.5, -0.25, 0 hours predose and at 1, 8, 24, 36, 48, 72, 96, 120, 144, 168, 240, 336 and 480 hours postdose.
Population: The analysis population included all participants randomized and treated who had at least 1 concentration in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 12 | 12
ng/mL | 8.834 (58) | 8.193 (51)

4. Primary Outcome: Corrected AUClast of Total Testosterone (Part 2).
Description: The AUClast of total testosterone in Part 2 of the study was observed directly from data. The baseline endogenous testosterone level was the mean of the 4 predose PK samples, an average baseline correction of endogenous total testosterone levels was calculated.
Time Frame: At -1, -0.5, -0.25, 0 hours predose and at 1, 8, 24, 36, 48, 72, 96, 120, 144, 168, 240, 336 and 480 hours postdose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 59 | 60
ng*hr/mL | 1251 (59) | 1384 (41)

5. Primary Outcome: Corrected AUCinf of Total Testosterone (Part 2).
Description: The AUCinf of total testosterone in Part 2 of the study was observed directly from data. The baseline endogenous testosterone level was the mean of the 4 predose PK samples, an average baseline correction of endogenous total testosterone levels was calculated.
Time Frame: At -1, -0.5, -0.25, 0 hours predose and at 1, 8, 24, 36, 48, 72, 96, 120, 144, 168, 240, 336 and 480 hours postdose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 43 | 50
ng*hr/mL | 1459 (44) | 1493 (40)

6. Primary Outcome: Corrected Cmax of Total Testosterone (Part 2)
Description: The Cmax of total testosterone in Part 2 of the study was observed directly from data. The baseline endogenous testosterone level was the mean of the 4 predose PK samples, an average baseline correction of endogenous total testosterone levels was calculated.
Time Frame: At -1, -0.5, -0.25, 0 hours predose and at 1, 8, 24, 36, 48, 72, 96, 120, 144, 168, 240, 336 and 480 hours postdose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 59 | 60
ng/mL | 8.891 (61) | 9.207 (50)

ADVERSE EVENTS:
Time Frame: From the signing of informed consent through and including a minimum of 28 calendar days and up to 35 calendar days after the last administration of the investigational product.
Description: Serious adverse events (SAEs) and non-serious AEs were recorded on the CRF. SAEs were also reported on the Clinical Trial (CT) SAE report form to Pfizer Safety within 24 hours of awareness.
Groups:
- Treatment A (Parts 1 and 2); Treatment B (Parts 1 and 2): This was a 2-part study, participants were enrolled in the 2 parts to receive Treatment A and Treatment B in different sequence. Treatment A (Test) was a single testosterone cypionate solution (new formulation) 200 mg dose administered for injection (IM) deep in the gluteal muscle. Treatment B (Reference) was a single testosterone cypionate solution for injection (currently marketed formulation) 200 mg administered IM deep in the gluteal muscle. This group included the participants enrolled in both Part 1 and Part 2 of the study.
Arm/Group | Treatment A (Parts 1 and 2) | Treatment B (Parts 1 and 2)
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72
Other Adverse Events (participants affected / at risk) | 7/71 | 1/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment A (Parts 1 and 2) (N=71) | Treatment B (Parts 1 and 2) (N=72)
Nasopharyngitis (Infections and infestations) | 4/59 | 0/60
Lip disorder (Gastrointestinal disorders) | 0/12 | 1/12
Skin Abrasion (Injury, poisoning and procedural complications) | 2/12 | 0/12
Alanine aminotransferase increased (Investigations) | 1/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03792477/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03792477/SAP_001.pdf